CLINICAL TRIAL: NCT03268096
Title: Disability, MRI Lesions and Thickness of Retinal Fibers: Evaluation 15 Years After a First Episode of Demyelination
Acronym: DB-SEP15
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: AGN_2017_6
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-02

CONDITIONS: Multiple Sclerosis; Pathologic Processes; Tomography, Optical Coherence; Magnetic Resonance Imaging; Prognosis
MeSH Terms: conditions — Multiple Sclerosis; Pathologic Processes | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Cerebral MRI and Optical Coherence Tomography — Clinical and paraclinical assessment (cerebral MRI and Optical Coherence Tomography) will be carried out on the same day. Paraclinical evaluation consists in the realization of additional MRI sequences in order to obtain more precise information on brain lesions (unconventional parameters). An optical coherence tomography will also be performed for both eyes to describe the thickness of the different layers of the retina.

SUMMARY:
Knowledge of the evolution of multiple sclerosis (MS) and its long-term prognostic factors is essential to guide the therapeutic management. However, it remains partial and concerns above all data collected during the first years of the disease. The evolution towards disability can only be assessed after a follow-up of more than 10 years and does not depend solely on the initial inflammatory activity of the disease. We propose to realize a standardized clinical assessment, an optical coherence tomography (OCT) and a cerebral MRI 15 years after the first clinical manifestation of the disease.

Clinical and paraclinical assessment will consist in the realization of additional MRI sequences in order to obtain more precise information on cerebral lesions (unconventional parameters). Optical coherence tomography (new generation device) will also be performed on both eyes to describe the thickness of the different layers of the retina. A clinical evaluation will be performed with the Expanded Disability Status Scale (EDSS).

This study aims:

1. to describe the current clinical situation of patients (e.g. percentage of patients with moderate or severe disability)
2. to explore the associations between MRI parameters, those measured with OCT and clinical characteristics (disability)
3. to explore clinical and paraclinical prognostic factors of pejorative evolution (disability, severe cerebral atrophy, etc.)

ELIGIBILITY:
Inclusion Criteria:

* First episode of demyelination occurred at least 10 years ago
* Hospitalized in the neurology department during this episode
* Insured with a social security scheme
* Having given his consent to participate in the study

Exclusion Criteria:

* Contraindications to 3 Tesla MRI and injection of contrast media
* Benefiting from a legal protection measure
* Pregnant or nursing mother

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had an episode of demyelination at least 10 years ago
Sampling Method: Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-03 (Actual)

PRIMARY OUTCOMES:
Disability assessed with EDSS (Expanded Disability Status Scale) | Baseline
  Disability assessment will be carried out using the EDS (Expanded Disability Status) Scale.
  This scale ranges from 0 to 10. Binary or ordered variables will be considered with various thresholds (for example, a score equal to 3 corresponds to moderate disorders ; a score equal to 6 corresponds to major disorders (need of a stick to walk 100 meters)).

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Guéguen, MD, Principal Investigator — Fondation Ophtalmologique A. de Rothschild
Locations (1):
- Fondation Ophtalmologique A. de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided